CLINICAL TRIAL: NCT04970199
Title: Cardiovascular Protective Role of Laser Acupuncture in Systemic Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P.T.REC/012/003252
Record Dates: First submitted 2021-07-11; First posted 2021-07-21 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: System; Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): thirty lupus women received laser acupuncture (active) for one month (3 days week) on acupoint number 14 of GV meridian, acupoint number 4 and 11 of large intestine, acupoint number 34 of gall bladder meridian, acupoint number 3 of liver meridian, acupoint number 4, 12, and 9 of conception vessel meridian, acupoint number 40, 36, and 25 of stomach meridian, acupoint number 6 of spleen meridian, and acupoint number 5 of triple energizer meridian (laser was applied for 1 min on every acupiont).
  Interventions: Device: laser application on acupoints
- group 2 (Sham Comparator): thirty lupus women received laser acupuncture (sham) for one month (3 days) on acupoint number 14 of GV meridian, acupoint number 4 and 11 of large intestine, acupoint number 34 of gall bladder meridian, acupoint number 3 of liver meridian, acupoint number 4, 12, and 9 of conception vessel meridian, acupoint number 40, 36, and 25 of stomach meridian, acupoint number 6 of spleen meridian, and acupoint number 5 of triple energizer meridian (laser was be applied for 1 min on every acupiont).
  Interventions: Device: laser application on acupoints

INTERVENTIONS:
Device: laser application on acupoints — laser acupuncture

SUMMARY:
Systemic lupus erythematosus is a chronic and multisystemic autoimmune disorder which predominantly affecting women. The most common cause of death in lupus patients affected by disease for more than 5 years is cardiovascular disease due to presence of some factors as oxidative stress, pro-inflammatory cytokines , dyslipidemia, diabetes, and hypertension.

DETAILED DESCRIPTION:
laser acupuncture (active or sham) for one month (3 days/week ) on acupoint number 14 of GV meridian, acupoint number 4 and 11 of large intestine, acupoint number 34 of gall bladder meridian, acupoint number 3 of liver meridian, acupoint number 4, 12, and 9 of conception vessel meridian, acupoint number 40, 36, and 25 of stomach meridian, acupoint number 6 of spleen meridian, and acupoint number 5 of triple energizer meridian (laser will be applied for 1 min on every acupiont) in lupus females

ELIGIBILITY:
Inclusion Criteria:

* lupus females
* 60 patients

Exclusion Criteria:

* pregnancy
* cardiovascular diseases
* respiratory diseases

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 60 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde | It was measured after 4 weeks
  anti-oxidative stress factor

SECONDARY OUTCOMES:
systole | It was measured after 4 weeks
  blood pressure
diastole | It was measured after 4 weeks
  blood pressure
blood glucose | It was be measured after 4 weeks
  fasting
erythrocyte sedimentation rate (1 hour) | It was measured after 4 weeks
  inflammatory marker
erythrocyte sedimentation rate (2 hour) | It was measured after 4 weeks
  inflammatory marker
c reactive protein | It was measured after 4 weeks
  inflammatory marker
adenosine triphosphate | It was measured after 4 weeks
  energy production marker
Nitrate | It was measured after 4 weeks
  oxidative stress factor
Glutathione | It was measured after 4 weeks
  antioxidant marker

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt